CLINICAL TRIAL: NCT07093450
Title: Estudo de Implementação de Melhoria de Qualidade Para Redução do Uso de Antimicrobianos em Unidades de Terapia Intensiva
Brief Title: Quality Improvement Intervention for a Safe Antimicrobial Use Reduction in Critically Ill Patients
Acronym: SAFE-REDUCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Collaborators: Hospital do Coracao (Other); Hospital Israelita Albert Einstein (Other); Beneficência Portuguesa de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 85063424.0.1001.5461
Record Dates: First submitted 2025-06-16; First posted 2025-07-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-07

CONDITIONS: Infection; Antimicrobial Stewardship; Critically Ill Intensive Care Unit Patients
Keywords: Antimicrobial stewardship; Intensive care unit; Infection; Stepped-wedge cluster trials; Hybrid effectiveness-implementation trials; Diagnostic stewardship
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: The study is a stepped-wedge cluster randomized trial, in which each of the 10 intensive care units will be randomized to receive a quality improvement intervention at each month. They will know about their allocation with 1-2 months preceding the commencement of the quality improvement intervention. There will be no transition period for the primary analysis. As the study is at the cluster level, no blinding will be possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICU Standard-of-care (No Intervention): The control group will be before the quality improvement intervention. Each ICU will be their own control and also the control group for ICUs that have already transitioned to the quality improvement arm.
  During this period, before transitioning to the educational QI intervention, ICUs will continue their routine standard-of-care, including any ongoing continuous quality improvement that takes part of the usual ICU management activities. Local ICUs have been disencouraged, though, to start any quality improvement initiatives aiming to improve antimicrobial consumption before their transition to the intervention phase.
- Educational Quality Improvement Intervention (Experimental): Participant ICUs who have transitioned to the quality improvement intervention will be part of this arm after their first visit. The intervention will consist of cognitive aids regarding antimicrobial initiation and duration for ICU physicians and healthcare professionals involved with antimicrobial decision-making. There will also be a monthly cross-sectional evaluation of the fidelity of the intervention, with immediate feedback at each assessment to the participating ICU.
  Interventions: Other: Educational Quality Improvement Intervention

INTERVENTIONS:
Other: Educational Quality Improvement Intervention — The intervention will be delivered at the cluster level. It will include an initiation visit, when educational sessions and an operations manual will be delivered to the ICU. These will consist of cognitive aids for antimicrobial initiation and duration decision-making, based on recent recommendations from guidelines, societies and regulatory authorities. In this visit, an assessment of barriers and facilitators for implementation of the behavioral change will be done, so that local adaptations can be done by the clinicians championing the implementation. Additionally, monthly, one-day audits will be done, which will be used to provide feedback to the ICU during the intervention phase regarding the suggested recommendations for antimicrobial decision-making.
  Arms: Educational Quality Improvement Intervention

SUMMARY:
The goal of this clinical trial is to learn if an educational intervention with audit and feedback on physicians and health care professionals who participate in antimicrobial treatment decisions can reduce the use of antimicrobials in adult patients admitted to a sample of Brazilian intensive care units (ICUs). The educational intervention is based on a literature review of current recommendations for a more rational use of antimicrobials and microbiological tests in daily ICU practice.

The main questions it aims to answer are:

* Does the educational intervention reduce the antimicrobial consumption in the intensive care units?
* Does this educational intervention aiming to reduce antimicrobial utilization in accordance with the latest guidelines have any safety signals regarding ICU mortality rates or ICU length-of-stay?

Researchers will compare (1) ICUs sequentially randomized to this quality improvement educational intervention aimed at improving antimicrobial utilization to (2) the same ICUs at months where the educational intervention has not been delivered yet.

Each participant ICU will transition to the quality improvement intervention approximately each month, starting at July, 2025. This quality improvement intervention is based on current recommendations for antimicrobial stewardship from regulatory agencies and medical societies, including cognitive aids for physicians to improve decision-making regarding the commencement of antimicrobials, their duration and antimicrobial time-outs. The investigators hypothesize that intensivists (ICU doctors) need to embrace antimicrobial stewardship as a core competence of their daily activities.

DETAILED DESCRIPTION:
The SAFE-REDUCE trial is a hybrid effectiveness-implementation type 1 trial, where the investigators intend to implement a quality improvement (QI) intervention aiming to improve antimicrobial utilization in a sample of intensive care units. Their hypothesis is that this QI intervention will reduce antimicrobial consumption in the studied intensive care units. For this implementation, due to logistical constraints, the investigators can only train one intensive care unit at a time and therefore they designed a stepped-wedge cluster randomized trial to evaluate the impact of this QI intervention.

The trial will be conducted in 10 intensive care units currently participating in the IMPACTO-MR platform, a registry focused on evaluating the impact of intensive care unit acquired infections and multidrug resistant infections. IMPACTO-MR routinely collects data from the participating ICUs, including standard ICU quality improvement data. Additionally, the platform collects data on antimicrobial utilization, reported ICU-acquired infections and microbiological culture results. In the SAFE-REDUCE trial, the investigators will take advantage of this ongoing registry to test if the educational QI intervention can modulate antimicrobial utilization while maintaining the trends of ICU mortality and length-of-stay.

Each participant ICU will go through a control phase, in which they will follow their current practice, and they will be transitioned to an intervention phase, in which the quality improvement intervention will be delivered to the intensive care unit.

The QI intervention will provide cognitive aids to ICU physicians aiming at improving their decision-making for antimicrobial initiation, antimicrobial time-outs (i.e, routine revisions of the actual need for antimicrobials) and, when an infection is highly likely, deciding appropriate, shorter durations of antimicrobials. The investigators will provide intensive care units with educational sessions, a written guide for antimicrobial initiation and duration decision-making, while also accounting for key diagnostic stewardship considerations. Following an initial site visit, the investigators will collect monthly point-prevalence surveys in the ICUs regarding antimicrobial utilization in one day of the month, for the duration of the trial. During these point-prevalence surveys, feedback will be provided to the ICU provider to be delivered to the ICU team. Additionally, during the first site visit, ICUs will be encouraged to evaluate barriers and facilitators to implement the educational intervention in their units, and they will be allowed to adapt further local training based on this assessment.

All participating ICUs of the SAFE-REDUCE stepped-wedge cluster randomized trial will be transitioned to the quality improvement intervention. The investigators included a baseline period (one month before implementation, expected on June, 2025, where only routinely collected data from the IMPACTO-MR platform will be linked to SAFE-REDUCE) in all ICUs and a phase-out phase (for three months, expected to occur on May-Jul, 2026) to evaluate whether any intervention benefits sustain after the investigators stop the point-prevalence surveys and feedback.

The investigators calculated sample size based on Hemming et al. suggested method. Considering that the study ICUs screened for participating in the SAFE-REDUCE trial would have between 10 and 30 ICU beds, most of them with 20 ICU beds, assuming a conservative occupation rate of 85%, the investigators estimated that 600 patient-days per period would be included, with each participating ICU transitioning to the intervention period in 10 steps. The investigators estimate the intervention will be able to reduce up to 20% the antimicrobial consumption in the ICU and they anticipate a variable baseline rate of antimicrobial utilization, considering an intracluster correlation coefficient (ICC) of 0.1. The investigators tested different ICCs, baseline daily defined doses and reductions in their level and the sample size yielded > 90% power in all simulations.

Given the analysis at the cluster level, informed consent was waived from the institutional review board at the coordinating center and at each participating hospital institutional review boards. They agreed with a minimal risk study (i.e., participation in this study will not incur higher risk than usual random variability observed in clinical practice) and the impossibility of obtaining informed consent to withdraw data utilization, as the primary outcome data is collected at the level of the unit, not at the level of the participants.

ELIGIBILITY:
Intensive care units inclusion Criteria:

* ICU leadership acceptance to participant in the quality improvement intervention;
* Hospital infection control leadership acceptance to participant in the quality improvement intervention;
* ICU participation in the IMPACTO-MR platform with high quality data;
* ICU potential for quality improvement based on a subjective assessment of the ICU and hospital infection leaderships

Intensive care units exclusion Criteria:

- Absence of local IRB approval

Participants inclusion Criteria:

* All patients admitted to the intensive care unit

Participants exclusion Criteria:

* Patients younger than 18 years-old will be excluded from individual-level analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9000 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Antimicrobial utilization at the ICU level | 14 months
  Antimicrobial utilization will be measured as daily defined doses (DDD) of antimicrobials at the ICU level per 100 patient-days

SECONDARY OUTCOMES:
ICU mortality rate | 14 months
  ICU mortality rate adjusted for illness severity at baseline (measured with the illness severity score SAPS 3)
ICU length-of-stay | 14 months
  ICU length-of-stay, adjusted for baseline illness severity (SAPS 3)

OTHER OUTCOMES:
Antimicrobial consumption, stratified by AWaRe WHO classification | 14 months
  Antimicrobial consumption measured as daily defined doses (DDDs) of antimicrobials, stratified by AWaRe WHO classification
Microbiological cultures collection rate | 14 months
  Microbiological cultures collection rate per patient-day. Results will be presented as a whole and stratified by sampling site (e.g., urinary, pulmonary, blood samples)
Microbiological cultures positivity rate | 14 months
  Microbiological cultures positivity rate per patient-day. Results will be presented as a whole and stratified by sampling site (e.g., urinary, pulmonary, blood samples)
Rate of skin-contaminant positive blood cultures | 14 months
  Skin-contaminant positive blood cultures rate per patient-day.
Resistance profile of positive microbiological isolates | 14 months
  Proportion of resistant microbiological isolates to important resistance phenotypes (for gram-negative: ceftriaxone resistance; carbapenem resistance; for gram-positive: oxacylin resistance and vancomycin resistance). Results will be presented as a whole and stratified by sampling site (e.g., urinary, pulmonary, blood samples) and type of bacteria (gram-positive or gram-negative; enterobacteria, Pseudomonas sp., Acinetobacter sp., others).
Ventilator-associated pneumonia (VAP) incidence rate | 14 months
  Ventilator-associated pneumonia (VAP) incidence rate, as reported by Brazilian regulatory agency criteria by local hospital infection control services.
Central-line associated bloodstream infection (CLABSI) incidence rate | 14 months
  Central-line associated bloodstream infection (CLABSI) incidence rate, as reported by Brazilian regulatory agency criteria by local hospital infection control services.
Catheter-associated urinary tract infection (CAUTI) incidence rate | 14 months
  Catheter-associated urinary tract infection (CAUTI) incidence rate, as reported by Brazilian regulatory agency criteria by local hospital infection control services.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno A M P Besen, M.D., Ph.D., Principal Investigator — Hospital Sírio-Libanês
Locations (9):
- Brazil (9):
  - Hospital Maternidade São José, Colatina, Espírito Santo
  - Santa Casa de Misericórdia de Passos, Passos, Minas Gerais
  - Hospital Municipal de Maringá, Maringá, Paraná
  - Hospital Pelópidas Silveira, Recife, Pernambuco
  - Hospital Naval Marcílio Dias, Rio de Janeiro, Rio de Janeiro
  - Hospital Onofre Lopes, Natal, Rio Grande do Norte
  - Hospital de Pronto Socorro, Porto Alegre, Rio Grande do Sul
  - Hospital Santa Cruz, Santa Cruz do Sul, Rio Grande do Sul
  - Santa Casa de Misericórdia de Barretos, Barretos, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data (IPD) might be shared upon request and approval by the study steering committee after the study completion.

REFERENCES:
- [Result] Tomazini BM, Nassar AP Jr, Lisboa TC, Azevedo LCP, Veiga VC, Catarino DGM, Fogazzi DV, Arns B, Piastrelli FT, Dietrich C, Negrelli KL, Jesuino IA, Reis LFL, Mattos RR, Pinheiro CCG, Luz MN, Spadoni CCDS, Moro EE, Bueno FR, Sampaio CSJC, Silva DP, Baldassare FP, Silva ACA, Veiga T, Barbante L, Lambauer M, Campos VB, Santos E, Santos RHN, Laranjeiras LN, Valeis N, Santucci E, Miranda TA, Patrocinio ACLD, Carvalho A, Sousa EMC, Sousa AHF, Malheiro DT, Bezerra IL, Rodrigues MB, Malicia JC, Silva SSD, Gimenes BDP, Sesin GP, Zavascki AP, Sganzerla D, Medeiros GS, Santos RDRMD, Silva FKR, Cheno MY, Abrahao CF, Oliveira Junior HA, Rocha LL, Nunes Neto PA, Pereira VC, Paciencia LEM, Bueno ES, Caser EB, Ribeiro LZ, Fernandes CCF, Garcia JM, Silva VFF, Santos AJD, Machado FR, Souza MA, Ferronato BR, Urbano HCA, Moreira DCA, Souza-Dantas VC, Duarte DM, Coelho J, Figueiredo RC, Foreque F, Romano TG, Cubos D, Spirale VM, Nogueira RS, Maia IS, Zandonai CL, Lovato WJ, Cerantola RB, Toledo TGP, Tomba PO, Almeida JR, Sanches LC, Pierini L, Cunha M, Sousa MT, Azevedo B, Dal-Pizzol F, Damasio DC, Bainy MP, Beduhn DAV, Jatoba JDVN, Moura MTF, Rego LRM, Silva AVD, Oliveira LP, Sodre Filho ES, Santos SSD, Neves IL, Leao VCA, Paes JLL, Silva MCM, Oliveira CD, Santiago RCB, Paranhos JLDR, Wiermann IGDS, Pedroso DFF, Sawada PY, Prestes RM, Nascimento GC, Grion CMC, Carrilho CMDM, Dantas RLAM, Silva EP, Silva ACD, Oliveira SMB, Golin NA, Tregnago R, Lima VP, Silva KGND, Boschi E, Buffon V, Machado AS, Capeletti L, Foernges RB, Carvalho AS, Oliveira Junior LC, Oliveira DC, Silva EM, Ribeiro J, Pereira FC, Salgado FB, Deutschendorf C, Silva CFD, Gobatto ALN, Oliveira CB, Dracoulakis MDA, Alvaia NOS, Souza RM, Araujo LLC, Melo RMV, Passos LCS, Vidal CFL, Rodrigues FLA, Kurtz P, Shinotsuka CR, Tavares MB, Santana IDV, Gavinho LMDS, Nascimento AB, Pereira AJ, Cavalcanti AB. IMPACTO-MR: a Brazilian nationwide platform study to assess infections and multidrug resistance in intensive care units. Rev Bras Ter Intensiva. 2022 Oct-Dec;34(4):418-425. doi: 10.5935/0103-507X.20220209-pt. Epub 2023 Mar 3. PMID 36888821